CLINICAL TRIAL: NCT04614415
Title: Multicenter, Double Blind, Randomized, Controlled Clinical Investigation to Evaluate the Performance of Autocross-linked Hyaluronic Acid for the Treatment of Hypertrophic Scars
Brief Title: Clinical Investigation to Evaluate the Performance of Hyaluronic Acid for the Treatment of Hypertrophic Scars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LQ5I-19-01
Record Dates: First submitted 2020-03-02; First posted 2020-11-04 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Hypertrophic Scar
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): group 1 will be treated with autocrosslinked Hyaluronic acid
  Interventions: Device: Autocrosslinked Hyaluronic aid
- control group (Placebo Comparator): group 2 treated with placebo (isotonic saline solution).
  Interventions: Other: placebo

INTERVENTIONS:
Device: Autocrosslinked Hyaluronic aid — IAL-SYSTEM ACP gel is an auto-cross-linked HA derivative in the form of highly viscous gel. In this direct formation of ester linkages no foreign substances are introduced into the molecule, thus catabolism of ACP leads only to HA
  Other Names: IAL SYSTEM ACP
  Arms: Treatment group
Other: placebo — The placebo consists in an isotonic saline solution (NaCl 0.9%)
  Arms: control group

SUMMARY:
The study includes two study groups, one involves treatment with auto-cross-linked Hyaluronic acid by intralesional and hypodermic injection, repeated after two weeks (T14), while the control arm provides an equal treatment but with isotonic saline solution.

Enrolled patients will be randomized into 2 groups with an allocation of 2:1 in study treatment arm and control arm respectively. They will be evaluated using the POSAS scale before the treatment and re-evaluated at 30, 90 and 180 days after treatment.

The scar evaluation will be completed by an ultrasound assessment at time 0 (T0), 30 (T30), T90 and T180 and the DLQI (Dermatology Life Quality Index) to be assessed at time 0 (T0), 30 (T30), 90 (T90) and 180 (T180).

In subjects that will consent, a small surgical biopsy for an explorative evaluation of the scar tissue will be performed before (T0) and after treatment (T30) for a histological assessment.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male or female subjects aged ≥ 18 and ≤ 85 years
* Subjects with hypertrophic scars caused by trauma, burn or iatrogenic injury with or without involvement of the mobile joints
* Scar > 2 to < 25 cm2 of surface
* Scar not previously treated with corticosteroids, laser or other invasive treatments
* Scar present for at least 12 months
* Scar located in all areas of the body with the exception of the face and neck
* Fitzpatrick skin score of I-VI
* Subjects willing to comply with all the steps of treatment and follow-up visits
* Subjects willing to refrain from any cosmetic intervention in the area to be treated during the clinical investigation
* Female of child-bearing potential (i.e. not in menopausal status from at least one year or permanently sterilized) must have a negative urine pregnancy test prior the first treatment

Exclusion Criteria:

Subjects with type I and type II diabetes mellitus

* Subjects with oncological diseases in progress or in remission
* Subjects receiving immunosuppressive drugs and corticosteroids, anticoagulants, antiplatelet agents
* Subjects with autoimmune diseases including connectivitis
* Subjects with congenital or acquired immunodeficiencies (including metabolic ones)
* Subjects with known allergy or hypersensitivity to hyaluronic acid or its derivatives
* Participation in clinical trials/investigations in the last 30 days
* Pregnant or breastfeeding women
* If female and of child-bearing potential, subject not using a highly effective method of birth control and not willing to use it during the participation to the clinical investigation
* Subjects not willing to avoid tanning during the clinical investigation
* Subjects with inflammations of the skin, including rosacea
* Subject with skin infection in the area to be treated
* Subjects having a high probability of non-compliance with the study procedures according to Investigator's judgement

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to Day 90 in POSAS total score for Observer | 90 days after treatment
  The performance of two injections of IAL-SYSTEM ACP in improving the quality of the scar after 90 days from the first treatment in patients with hypertrophic scars will be evaluated by the mean change from baseline to Day 90 in POSAS total score for Observer.

SECONDARY OUTCOMES:
To evaluate the performance of IAL-SYSTEM ACP in improving the quality of the scar | after 30 and 180 days from the first treatment
  Change from baseline to post-baseline visits (T30, T90 and T180) in total POSAS scores (sum total of Patient and Observer scores), and POSAS total score for Patient and Observer
To assess the changing in the Quality of life after 30, 90 and 180 days from the first treatment with the Dermatology Life Quality Index (DLQI) | after 30, 90 and 180 days from the first treatment
  Change from baseline to post-baseline visits (T30, T90 and T180) in DLQI score (dermatology quality of life Index)
To assess the changing in the dermal volume after 30, 90 and 180 days from the first treatment | after 30, 90 and 180 days
  Change from baseline to post-baseline visits (T30, T90 and T180) in dermal volume measured by ultrasound
Safety of the treatment. Number of patients with treatment related adverse events | throug clinical investigation completion, an average one year
  Safety evaluation examining the local and systemic adverse effects as consequence of the treatment and any other adverse event occurred during the study.

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - AOU Ospedali Riuniti- SOD Chirurgia ricostruttiva e chirurgia della mano, Ancona
  - U.O. Centro Grandi Ustionati Ospedale Bufalini di Cesena - AUSL, Cesena
  - U.O.C. Chirurgia Plastica e Centro Ustioni Azienda Ospedaliero-Universitaria di Parma, Parma
  - U.O.C. Centro Ustioni Azienda Ospedaliero-Universitaria Pisana, Pisa

IPD SHARING:
Plan to Share IPD: No